CLINICAL TRIAL: NCT04734379
Title: A Phase 2a Open-Label Preliminary Safety, Tolerability, and Biomarker Study of Oral Fasudil in Patients With the 4-Repeat Tauopathies of Progressive Supranuclear Palsy-Richardson Syndrome or Corticobasal Syndrome.
Brief Title: Rho Kinase (ROCK) Inhibitor in Tauopathies - 1
Acronym: ROCKIT-1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Woolsey Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WP-0512-002
Record Dates: First submitted 2021-01-18; First posted 2021-02-02 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Progressive Supranuclear Palsy; Corticobasal Syndrome
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Corticobasal Degeneration | interventions — fasudil

STUDY DESIGN:
Intervention Model Description: Open label, single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Oral fasudil 180 mg/day
  Interventions: Drug: Fasudil

INTERVENTIONS:
Drug: Fasudil — Oral fasudil 180 mg/day

SUMMARY:
A Phase 2a Open-Label Preliminary Safety, Tolerability, and Biomarker Study of Oral Fasudil in Patients with the 4-Repeat Tauopathies of Progressive Supranuclear Palsy-Richardson Syndrome or Corticobasal Syndrome

DETAILED DESCRIPTION:
After consent, participants will undergo screening evaluations, which may occur over the course of up to 6 weeks. Subjects who meet inclusion/exclusion criteria will be enrolled into the study and complete baseline evaluations. Dosing with study drug will begin on Day 1 and continue for 48 weeks. Participants will return to the clinic at Week 1 (7 ± 2 days after the first study drug administration) and at Weeks 12, 24, 36, and 48 for study evaluations, and at Week 52 for post-treatment follow-up evaluations. Plasma biomarker collection will occur at baseline, and Weeks 12, 24, 36, and 48. Cerebrospinal fluid (CSF) Biomarker collection will occur at screening, Week 24 and Week 48. Brain magnetic resonance imaging (MRI) will occur at screening, and Weeks 24 and 48. Safety labs will be collected at each study visit as well as during Week 4.

Adverse events (AEs) will be assessed at all visits and subjects will be contacted one day after the start of treatment (that is, one day after Visit 1), and monthly thereafter including at each visit. Subject will also be contacted one day after Visit 6/last day of dosing with study drug for subjects who discontinue early.

Subjects/caregivers will be queried for study drug compliance one day after the start of treatment (that is, one day after Visit 1), and monthly thereafter.

After completion of the 48-week primary portion of the study, subjects will be given the option to continue open-label treatment for up to an additional 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Between 35 and 80 years of age (inclusive).
2. Able to walk at least 10 steps with minimal assistance (stabilization of one arm or use of cane/walker).
3. MRI at Screening is consistent with the underlying neurodegenerative disease of the respective diagnostic cohort (i.e. PSP-RS or CBS), with no large strokes or severe white matter disease.
4. Mini-Mental State Exam (MMSE) at Screening is between 20 and 30 (inclusive).
5. For CBS: Amyloid beta (Aβ) positron emission tomography (PET) scan (florbetapir or equivalent) at Screening is not consistent with underlying Alzheimer's disease (AD). Previous Aβ PET scan negativity (assessed by a certified neuroradiologist) or previous AD CSF biomarker (Aβ/tau level, P-tau181 or Aβ1-40 / Aβ1-42) or plasma AD biomarker (P-tau181 or P-tau217) negativity may be used instead of performing an Aβ PET scan at Screening at the Principal Investigator's (PI's) discretion.
6. The following medications are allowed, but must be stable for 2 months prior to Baseline:

   1. FDA-approved AD medications
   2. FDA-approved Parkinson's Disease (PD) medications
7. Other prescription medications are allowed as long as the dose is stable for 30 days prior to Baseline. (Note Exclusion Criteria 17 and 18.)
8. Has a reliable study partner who agrees to accompany the participant to visits, and spends at least 5 hours per week with the participant.
9. Signed and dated written informed consent obtained from the participant/legally authorized representative (LAR) and the participant's study partner in accordance with local Institutional Review Board (IRB) regulations.
10. Women of childbearing potential (WCBP) must agree to abstain from sex or use an adequate method of contraception for the duration of the screening period, the study drug treatment period, and for 28 days after the last dose of study drug.
11. Males must agree to abstain from sex with WCBP or use an adequate method of contraception for the duration of the study drug treatment period and for 75 days after.

    For PSP-RS Only
12. Meets 2017 consensus criteria for possible or probable progressive supranuclear palsy-Richardson syndrome (PSP-RS).

    For CBS Only
13. Meets 2013 consensus criteria for possible or probable corticobasal degeneration (CBD), CBS subtype.

Exclusion Criteria:

1. Meets criteria for probable AD established by the National Institute on Aging and the Alzheimer's Association (NIA-AA).
2. Any other medical condition other than PSP-RS or CBS that could account for cognitive or motor deficits (e.g., active seizure disorder, stroke, vascular dementia, substance abuse or alcoholism).
3. History of a prominent and sustained response to levodopa therapy in the opinion of the PI.
4. Presence of significant cardiovascular, hematologic, renal, or hepatic disease.
5. Suicidal ideation per the Columbia-Suicide Severity Rating Scale (C-SSRS) that in the opinion of the PI would pose a safety risk or interfere with the appropriate interpretation of study data
6. History of major psychiatric illness or untreated depression that in the opinion of the PI would pose a safety risk or interfere with the appropriate interpretation of study data.
7. Neutrophil count <1,500/mm3, platelets <100,000/mm3, total bilirubin ≥1.5 x Upper Limit of Normal (ULN), alanine aminotransferase (ALT) ≥3 x ULN, aspartate aminotransferase (AST) ≥3 x ULN, or International Normalized Ratio (INR) >1.2.
8. Serum creatinine >1.3 mg/dL.
9. Evidence of any clinically significant findings on screening or baseline evaluations which, in the opinion of the PI would pose a safety risk or interfere with appropriate interpretation of study data.
10. Current or recent history (within four weeks prior to Screening) of a clinically significant bacterial, fungal, or mycobacterial infection.
11. Current clinically significant viral infection.
12. Major surgery within four weeks prior to Screening.
13. Any contraindication for MRI or unable to tolerate MRI scan at Screening.
14. Any contraindication to or unable to tolerate lumbar puncture at Screening, including use of anticoagulant medications such as warfarin. Daily administration of aspirin up to 81mg is not a contraindication, as long as the dose is stable for 30 days prior to Screening.
15. Participants who, in the opinion of the PI, are unable or unlikely to comply with the dosing schedule or study evaluations.
16. Treatment with another investigational drug within 30 days or 5 half-lives of drug before Baseline, whichever is longer. Treatment with investigational drugs other than fasudil while on study will not be allowed.
17. Treatment with systemic corticosteroids within 30 days or 5 half-lives of drug before Baseline, whichever is longer.
18. On more than one of the following drug classes: long-acting nitrates, beta-blockers, or calcium channel blockers.
19. Known hypersensitivity to the inactive ingredients in the study drug (fasudil).
20. Known to be pregnant or lactating; or positive pregnancy test at Screening or Baseline (Day 1) for WCBP.
21. Cancer within 5 years of Screening, except for basal cell carcinoma.
22. History of serum or plasma progranulin level less than one standard deviation below the normal participant mean for the laboratory performing the assay.
23. History or evidence at Screening of known disease-associated mutations in GRN, TBK1, C9ORF72, TARBP, CHMPB2, or VCP genes (FTLD causative gene mutations not associated with underlying tau pathology).
24. Blood pressure < 90/60.
25. Evidence of orthostatic hypotension.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 48 weeks
  Incidence of adverse events [AEs] and serious adverse events [SAEs] as assessed by clinically significant abnormal physical examination findings; changes in vital signs; 12-lead electrocardiogram [ECG]; magnetic resonance imaging [MRI]; and hematology, blood chemistry, liver function, and urine tests.

SECONDARY OUTCOMES:
Phosphorylated tau | 48 weeks
  Number of participants with changes in concentrations of cerebrospinal fluid (CSF) and plasma phosphorylated tau
Biomarkers of neurodegeneration | 48 weeks
  Number of participants with changes in biomarkers of neurodegeneration, including neurofilament light chain (NfL), and total tau fragment levels.
Imaging biomarkers of neurodegeneration | 48 weeks
  Number of participants with changes in imaging biomarkers of neurodegeneration, including changes in brain volume (whole brain, ventricles, hippocampus, frontal operculum, pre-central gyri, midbrain, pons and superior cerebellar peduncle) and white matter tract integrity (aslant tract, superior longitudinal fasciculus, and superior cerebellar peduncle) as determined by T1-weighted volumetric magnetic resonance imaging (MRI), diffusion tensor imaging (DTI)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ljubenkov, MD, Principal Investigator — UCSF Weill Institute for Neurosciences
Locations (1):
- University of California Weill Institute for Neurosciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No